CLINICAL TRIAL: NCT02912598
Title: Lung Isolation in Thoracic Surgery - a Comparison of the VivaSight™ EB Endobronchial Blocker With Established Devices
Brief Title: Lung Isolation in Thoracic Surgery - a Randomized Trial Comparing the VivaSight™ EB Endobronchial Blocker With Established Devices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Tom Kreft, Principal Investigator, Otto-von-Guericke University Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 142/14
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Lung Separation Techniques; One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mallinckrodt™ Endobronchial Tube (Active Comparator): Usage of a left-sided Mallinckrodt™ double-lumen tube (DLT) to achieve lung isolation and one lung ventilation.
  Interventions: Device: Mallinckrodt™ Endobronchial Tube
- Fuji Uniblocker™ (Active Comparator): Usage of a Fuji Uniblocker™ in a generic single-lumen tube to achieve lung isolation and one lung ventilation.
  Interventions: Device: Fuji Uniblocker™
- ETView VivaSight™-SL+EB (Experimental): Usage of a ETView VivaSight™-EB endobronchial blocker in a ETView VivaSight™-SL single-lumen tube to achieve lung isolation and one lung ventilation.
  Interventions: Device: ETView VivaSight™-SL+EB
- COOK© Arndt Endobronchial Blocker (Active Comparator): Usage of a COOK© Arndt Endobronchial Blocker in a generic single-lumen tube to achieve lung isolation and one lung ventilation.
  Interventions: Device: COOK© Arndt Endobronchial Blocker

INTERVENTIONS:
Device: Mallinckrodt™ Endobronchial Tube
  Arms: Mallinckrodt™ Endobronchial Tube
Device: Fuji Uniblocker™
  Arms: Fuji Uniblocker™
Device: ETView VivaSight™-SL+EB
  Arms: ETView VivaSight™-SL+EB
Device: COOK© Arndt Endobronchial Blocker
  Arms: COOK© Arndt Endobronchial Blocker

SUMMARY:
Surgery involving the chest cavity, particularly VATS procedures, often require one-lung ventilation. The double-lumen tube (DLT) is considered the gold standard for lung isolation with different models of bronchial blockers (BB) used in special populations and circumstances. Their routine use is impeded by prolonged placement times, frequent malpositionings and higher costs when compared to the DLT, as recently reported in a meta-analysis by Clayton-Smith et al. The VivaSight™ SL+EB as a combination of a single-lumen tube with an integrated camera and a bronchial blocker allows for endobronchial placement without the use of a fiberoptic bronchoscope. An external monitor provides continuous visualization of the tracheal carina and the position of the bronchial cuff. The purpose of this study was to evaluate the clinical performance of the VivaSight™ SL+EB when compared to a left-sided double-lumen tube and established bronchial blockers. The investigators hypothesized a reduction in time to initial lung isolation due to the simplified placement procedure compared to other bronchial blockers. Continuous intraprocedural airway visualization may allow for early detection of dislocations. Necessary repositionings may be possible without additional bronchoscopies, reducing both disruptions of ventilation and maintenance costs.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or at 18 years
* scheduled for elective thoracic surgery with one-lung ventilation
* written informed consent in anaesthesia, the study and anonymized data collection

Exclusion Criteria:

* necessary conversion between devices
* one-lung ventilation impossible to establish
* denial of the study or data collection
* surgical or anatomical circumstances preventing the use of a double-lumen tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to initial lung isolation | intraoperative
  Duration of initial bronchoscopy-guided placement of the endobronchial ballon. Start: Beginning of direct laryngoscopy. End: Initial inflation of the endobronchially placed cuff.

SECONDARY OUTCOMES:
Ease of placement [numerical rating scale] | intraoperative
  Evaluation of difficulty of endobronchial device placement by the anaesthetist.
Rate of dislocation | intraoperative
  Number of device dislocations after correct initial placement. Measurement time point after termination of one-lung ventilation.
Quality of surgical exposure [numerical rating scale] | intraoperative
  Surgeon's grading of the quality of surgical exposure resulting from lung deflation. Time point is initial view of the thoracic cavity after pleural incision.
Oxygenation | intraoperative
  Measurement of arterial partial pressure of oxygen by blood gas analysis taken 5min and 15min after establishment of one-lung ventilation.
Bronchoscopies | intraoperative
  Number of additional bronchoscopies required after initial placement resulting from suspected or actual dislocations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hachenberg, Prof. Dr. med., Study Chair — Klinik für Anaesthesiologie und Intensivtherapie der Otto-von-Guericke-Universität / Medizinische Fakultät Universitätsklinikum Magdeburg A.ö.R.